CLINICAL TRIAL: NCT00237328
Title: The Incidence of Thromboembolic Events in Patients With Antibodies to Heparin-PF4 After Cardiac Bypass
Brief Title: Risk of Developing Antibodies to Heparin-PF4 After Heart Surgery
Acronym: HIT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00010736
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Thrombosis
Keywords: Heparin resistance; Blood clotting; Heart surgery; Cardiopulmonary bypass
MeSH Terms: conditions — Thrombosis | interventions — Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Heparin — Heparin will be used as the intra-operative anticoagulant

SUMMARY:
Heparin is a drug that is widely used to prevent and treat blood clotting. Individuals undergoing cardiopulmonary bypass surgery are administered high doses of heparin, and some of them develop antibodies to the drug. This immune response can lead to the formation of blood clots, setting the stage for a potential heart attack or stroke. The purpose of this study is to evaluate how often an immune response to heparin leads to the formation of blood clots in individuals who have had heart surgery.

DETAILED DESCRIPTION:
Heparin is a drug that is widely used to prevent and treat blood clotting. However, heparin can also cause serious adverse events. Individuals undergoing cardiopulmonary bypass surgery are administered and therefore exposed to high doses of heparin. Studies have shown that up to 61% of cardiac bypass patients develop elevated levels of antibodies to heparin-PF4 after surgery. This immune response may activate blood platelets, possibly resulting in a blood clot. These clots most often develop in the legs and lungs, and may lead to a heart attack or stroke. The frequency of such a reaction has yet to be determined definitively. This study will evaluate the incidence of an immune response to heparin-PF4 that leads to the formation of blood clots in individuals who have had heart surgery.

Participants in this study will be recruited prior to a scheduled cardiac bypass surgery. They will first complete a structured pre-operative interview to collect baseline measures on demographics, comorbidities, history of heparin exposures, and prior thromboembolic events. Immediately prior to surgery, a blood sample will be taken to assess the individual's platelet count and level of antibodies to heparin-PF4. Following the operation, participants will be followed daily to assess heparin exposure, platelet counts, and any blood clotting. Subsequent blood samples will be taken 5 days and 1 month following the surgery to again evaluate the individual's platelet count and level of heparin-PF4 antibodies. Additionally, participants will undergo a structured interview at 1 and 3 months post-surgery to evaluate the incidence of outcomes related to heparin-PF4 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cardiac bypass surgery at Duke University Hospital

Exclusion Criteria:

* Plans to receive warfarin during the post-operative inpatient stay
* Plans to receive a full anticoagulant dose of low-molecular weight heparin during the post-operative inpatient stay
* Plans to receive a full anticoagulant dose of unfractionated heparin during the post-operative inpatient stay
* Use of any drug other than unfractionated heparin for anticoagulation during cardiopulmonary bypass
* Warfarin, heparin, or low-molecular weight heparin administered during a readmission to the hospital for a reason other than one of this study's outcomes does not constitute criteria for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing cardiac bypass surgery with heparin as the intra-operative anticoagulant at Duke University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Thrombotic events compatible with HIT | one year

SECONDARY OUTCOMES:
antibody positibe status post operative day 5 and day 30 | one year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ortel, MD, PhD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Warkentin TE, Greinacher A. Heparin-induced thrombocytopenia: recognition, treatment, and prevention: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):311S-337S. doi: 10.1378/chest.126.3_suppl.311S. PMID 15383477
- [Background] Alsoufi B, Boshkov LK, Kirby A, Ibsen L, Dower N, Shen I, Ungerleider R. Heparin-induced thrombocytopenia (HIT) in pediatric cardiac surgery: an emerging cause of morbidity and mortality. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2004;7:155-71. doi: 10.1053/j.pcsu.2004.02.024. PMID 15283365
- [Background] Pouplard C, May MA, Iochmann S, Amiral J, Vissac AM, Marchand M, Gruel Y. Antibodies to platelet factor 4-heparin after cardiopulmonary bypass in patients anticoagulated with unfractionated heparin or a low-molecular-weight heparin : clinical implications for heparin-induced thrombocytopenia. Circulation. 1999 May 18;99(19):2530-6. doi: 10.1161/01.cir.99.19.2530. PMID 10330384
- [Background] Warkentin TE, Greinacher A. Heparin-induced thrombocytopenia and cardiac surgery. Ann Thorac Surg. 2003 Dec;76(6):2121-31. doi: 10.1016/j.athoracsur.2003.09.034. PMID 14667668
- [Background] Williams RT, Damaraju LV, Mascelli MA, Barnathan ES, Califf RM, Simoons ML, Deliargyris EN, Sane DC. Anti-platelet factor 4/heparin antibodies: an independent predictor of 30-day myocardial infarction after acute coronary ischemic syndromes. Circulation. 2003 May 13;107(18):2307-12. doi: 10.1161/01.CIR.0000066696.57519.AF. Epub 2003 Apr 21. PMID 12707235